CLINICAL TRIAL: NCT01808716
Title: Effect of Low-level Laser Therapy (808nm) on Marker of Muscle Damage: Randomized Double-blind Placebo-controlled Study
Brief Title: Effect of Low-level Laser Therapy (808nm) on Marker of Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Cleber Ferraresi, Cleber Ferraresi, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP/UFRN 176/10
Record Dates: First submitted 2013-03-01; First posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: low-level laser therapy; muscle damage
MeSH Terms: interventions — Low-Level Light Therapy; Exercise Therapy; Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Low-level laser therapy (LLLT) on muscle damage (Active Comparator): Effects of low-level laser therapy (LLLT)on muscle damage
  Interventions: Device: Low-level laser therapy (808nm) and exercise
- Low-level laser therapy (LLLT) placebo on muscle damage (Active Comparator): Effects of low-level laser therapy (LLLT) placebo on muscle damage
  Interventions: Device: Low-level laser therapy (808nm) and exercise

INTERVENTIONS:
Device: Low-level laser therapy (808nm) and exercise — Use of low-level laser therapy(LLLT)or placebo-LLLT applied on biceps brachii for muscle damage recovery
  Other Names: Laser device (808nm; 100mW; DMC®, Brazil); Low-level laser therapy; Muscle damage; Muscle recovery

SUMMARY:
The study hypothesis is a decreased muscle damage induced by exercises when low-level laser therapy is applied on body muscles before exercises.

DETAILED DESCRIPTION:
The study assessed males submitted to exercise to induce muscle damage. Creatine kinase levels in blood was quantified in order to identify the magnitude of muscle damage.

ELIGIBILITY:
Inclusion Criteria:

* healthy males,
* physically active,
* aged between 25-40 years.

Exclusion Criteria:

* smoker, or
* under medicine as anti-inflammatory and/or any drug that could affect normal and physiological conditions and lesion in upper limbs.

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Creatine Kinase analysis in blood | 72 hours
  Evaluation of Creatine Kinase (CK) levels in blood before, immediately after and 24h, 48h and 72h after protocol of exercise to induce muscle damage

CONTACTS AND LOCATIONS:
Overall Officials: Wouber Hérickson de Brito Vieira, PhD, Study Director — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal Univesity of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

REFERENCES:
- [Background] Vieira WH, Ferraresi C, Perez SE, Baldissera V, Parizotto NA. Effects of low-level laser therapy (808 nm) on isokinetic muscle performance of young women submitted to endurance training: a randomized controlled clinical trial. Lasers Med Sci. 2012 Mar;27(2):497-504. doi: 10.1007/s10103-011-0984-0. Epub 2011 Aug 26. PMID 21870127
- [Background] Ferraresi C, de Brito Oliveira T, de Oliveira Zafalon L, de Menezes Reiff RB, Baldissera V, de Andrade Perez SE, Matheucci Junior E, Parizotto NA. Effects of low level laser therapy (808 nm) on physical strength training in humans. Lasers Med Sci. 2011 May;26(3):349-58. doi: 10.1007/s10103-010-0855-0. Epub 2010 Nov 18. PMID 21086010